CLINICAL TRIAL: NCT06129708
Title: Effect of Aquatic Exercise Versus Aerobic Exercise on Primary Dysmenorrhea and Quality of Life in Adolescent Females: A Randomized Controlled Trial
Brief Title: Effect of Aquatic Exercise Versus Aerobic Exercise on Primary Dysmenorrhea and Quality of Life in Adolescent Females
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Asmaa Yossry Abdelrahman Ahmed, Physical Therapist at Shubra General Hospital, PhD student at Department of Physical Therapy for Women's Health, Faculty of Physical Therapy, Cairo University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/004770
Record Dates: First submitted 2023-11-08; First posted 2023-11-13 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Dysmenorrhea Primary
Keywords: Primary Dysmenorrhea; Adolescent Females; Aquatic Exercise; Aerobic Exercise; Pressure Pain Threshold; Quality of Life
MeSH Terms: interventions — Aquatic Therapy; Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group (A) Aquatic Exercise Group (Experimental): They participated in an aqua aerobic exercise program, 3 days per week, for 8 weeks
  Interventions: Other: Aquatic Exercise
- Group (B) Aerobic Exercise Group (Experimental): They participated in an aerobic exercise program on a treadmill, 3 days per week, for 8 weeks.
  Interventions: Other: Aerobic Exercise

INTERVENTIONS:
Other: Aquatic Exercise — The aquatic exercises included 5 minutes of warming up in form of walking and running in water, 20 minutes of aerobic and strengthening exercises of pelvis, abdominal and thigh muscles (Double-leg Squat, lunge, knee flexion and extension, hip flexion and
  Arms: Group (A) Aquatic Exercise Group
Other: Aerobic Exercise — The exercise protocol consists of 5 minute warm up, 35 min aerobic exercise and 5 minute cool-down. Exercises high-intensity treadmill-based treatment for primary dysmenorrhea for three days a week ,The Borg Rating of Perceived Exertion (RPE) Scale from 6 ('no exertion at all') to 20 ('maximal exertion') was used to regulate the exercise intensity on the treadmill. Participants were encouraged to increase the speed of the treadmill until they perceived their RPE to be between 14 and 16. or at a perceived exertion of 11.0 (Borg scale) for the first five minutes (warm-up period), followed by aerobic exercise at 70-85% of maximum heart rate (MHR) (16.0-18.0 Borg scale) for 30 minutes. At the end of the exercise session, women completed a 5-minute cool-down (11.0 Borg scale).
  Arms: Group (B) Aerobic Exercise Group

SUMMARY:
This study was conducted to determine the difference between impact of aerobic and aquatic exercise on primary dysmenorrhea and quality of life in adolescent girls.

DETAILED DESCRIPTION:
Dysmenorrhea manifests as painful menstrual flow it occurs in two forms primary and secondary. Primary and secondary dysmenorrhea is painful menstruation occur without any gynecological disease it was conducted that prevalence of dysmenorrhea 74.6% and it was significantly more frequent in students from rural residence (Shaimaa et al., 2018).

There is only one previous study investigate effect of aquatic exercise on primary dysmenorrhea (Rezvani et al., 2013). There are several previous studies investigate effect of aerobic ex , however non of the previous studies compared between effect of aerobic and aquatic exercise on primary dysmenorrhea and quality of life of adolescent girls .Therefore this study was the first one which aimed to investigate the difference between effect of aerobic and aquatic exercise on primary dysmenorrhea and quality of life in adolescent girls.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, nonsmoking, virginal girls having moderate to severe primary dysmenorrhea (score on pain rating scale > 3).
* Their ages ranged from 14 to 20 years
* Their body mass index (BMI) ranged from 18 to 25 kg/m2.
* They haven't practice any sports at least one year

Exclusion Criteria:

* Any musculoskeletal disorder.
* Cardio-respiratory disease.
* Diabetes, hypertension, or anemia.
* Adolescent girls who have utilized hormonal treatment in the six months prior to study commencement.
* currently undergoing pharmacological therapy for menstrual pain management

Ages: 14 Years to 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 60 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
Assessment of dysmenorrhea severity | 12 weeks
  It was assessed for each participant in the two groups (A & B) before and after 12 weeks of treatment at the first day of menstruation, using WaLIDD scale, which has high sensitivity and high specificity.
Measurement of pain intensity | 12 weeks
  It was measured for each participant in both groups (A & B) before and after 12 weeks of treatment at the first day of menstruation, using the Arabic version of numeric pain rating scale. The respondents were required to select a number (0-10 integers) that best reflected the intensity of her pain. In the numeric pain rating scale, 0 represented no pain, 1-3 indicated mild pain, 4-6 indicated moderate pain, while 7-10 indicated severe pain.
Assessment of pressure pain threshold (PPT) | 12 weeks
  The PPT was measured for each participant in both groups (A & B) before and after 12 weeks of treatment at the first day of menstruation, using a pressure algometry.
Assessment of health related quality of life | 12 weeks
  The health related quality of life of all participants in both groups (A & B) was evaluated before and after the end of treatment program, using the Arabic version of EQ-5D-3L questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Sohier M. Elkosery, Prof., Study Chair — Department of Physical Therapy for Woman's Health, Faculty of physical therapy, Cairo University, Giza, Egypt.
Locations (1):
- Cairo University, Giza, Egypt

REFERENCES:
- [Derived] Abdelrahman AY, El-Kosery SM, Abbassy AH, Botla AM. Effect of aquatic exercise versus aerobic exercise on primary dysmenorrhea and quality of life in adolescent females: A randomized controlled trial. Physiother Res Int. 2024 Jul;29(3):e2095. doi: 10.1002/pri.2095. PMID 38767193